CLINICAL TRIAL: NCT00004202
Title: A Phase II Study of Induction Chemotherapy With Paclitaxel and Carboplatin Followed by Radiation Therapy With RSR13 for Locally Advanced Inoperable Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy, Radiation Therapy, and RSR13 in Treating Patients With Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067445; ALLOS-RSR13RT-010; VU-VCC-THO-9828
Record Dates: First submitted 2000-01-21; First posted 2004-06-25 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Drug Therapy; efaproxiral; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: chemotherapy
Drug: efaproxiral
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as RSR13 may make tumor cells more sensitive to radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, radiation therapy, and RSR13 in treating patients who have stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the one year survival rate, two year survival rate, and median survival rate in patients with locally advanced unresectable non-small cell lung cancer treated with paclitaxel and carboplatin followed by radiotherapy plus RSR13. II. Determine the complete and partial response rates and progression free interval in the chest (radiation portal) of these patients on this regimen. III. Determine the time to disease progression outside of the radiation portal in these patients on this regimen. IV. Determine the toxic effects and adverse events associated with this regimen in these patients.

OUTLINE: This is a multicenter study. Induction chemotherapy: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes every 3 weeks for 2 courses. Radiotherapy: Beginning 3 to 4 weeks after induction chemotherapy, patients receive RSR13 IV over 30 minutes, followed by fractionated radiotherapy 5 times weekly for 6-7 weeks. Patients are followed monthly for 2 months and then every 3 months thereafter until disease progression or death.

PROJECTED ACCRUAL: A total of 46-48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally advanced unresectable stage IIIA or IIIB non-small cell lung cancer (NSCLC), including: Squamous cell carcinoma OR Adenocarcinoma (including bronchoalveolar cell) OR Large cell anaplastic carcinoma (including giant and clear cell) OR Poorly differentiated NSCLC No small cell carcinoma No distant metastases Measurable or evaluable disease by chest x-ray, CT, or MRI scan Tumors adjacent to vertebral body are eligible if all gross disease is in the radiation boost field No pleural effusion(s) that are exudative, bloody, or cytologically malignant No asymptomatic brain metastases by CT or MRI scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL (transfusion or epoetin alfa allowed) Hepatic: Bilirubin less than 1.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: No uncontrolled serious cardiac disease No active congestive heart failure, unstable angina, pericardial effusion, or arrhythmia Pulmonary: FVC or FEV1 at least 50% Resting or exercise SaO2 on room air at least 90% by pulse oximetry Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active concurrent malignancy within the past 5 years, except: Nonmelanomatous skin cancer Carcinoma in situ of the cervix No serious medical or psychiatric illness that would preclude compliance No active serious infection No concurrent clinically significant peripheral neuropathy No prior significant allergic reaction to drugs containing Cremophor (e.g., cyclosporine or vitamin K) No greater than 10% weight loss in the past 3 months

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic therapy No concurrent immunotherapy (during radiotherapy (RT) and RSR13 administration) Chemotherapy: No prior systemic chemotherapy No concurrent chemotherapy (during RT and RSR13 administration) Endocrine therapy: No concurrent hormonal therapy (during RT and RSR13 administration) Radiotherapy: No prior radiotherapy to the thorax Surgery: At least 1 week since prior diagnostic thoracoscopy OR At least 3 weeks since prior thoracotomy and recovered No prior total surgical resection Other: At least 3 weeks since other prior investigational agents or devices No prior RSR13

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-10 (Actual); Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hak Choy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (16):
- United States (10):
  - Arizona Cancer Center, Tucson, Arizona
  - Cedars-Sinai Comprehensive Cancer Center, Los Angeles, California
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Cancer Center of Albany Medical Center, Albany, New York
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Boston Cancer Group, Memphis, Tennessee
  - Dan Rudy Cancer Center, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Massey Cancer Center, Richmond, Virginia
- Canada (6):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Centre Universitaire de Sante de l'Estrie - Site Fleurimont, Fleurimont, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Notre Dame Hospital, Montreal, Quebec

REFERENCES:
- [Background] Choy H, Swann S, Nabid A, et al.: Comparison of 5-year survival between RTOG-94-10 and a phase 2 study of induction chemotherapy followed by efaproxiral + radiotherapy in patients with locally advanced NSCLC. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-49, S28-9, 2006.
- [Result] Choy H, Nabid A, Stea B, Scott C, Roa W, Kleinberg L, Ayoub J, Smith C, Souhami L, Hamburg S, Spanos W, Kreisman H, Boyd AP, Cagnoni PJ, Curran WJ. Phase II multicenter study of induction chemotherapy followed by concurrent efaproxiral (RSR13) and thoracic radiotherapy for patients with locally advanced non-small-cell lung cancer. J Clin Oncol. 2005 Sep 1;23(25):5918-28. doi: 10.1200/JCO.2005.08.011. PMID 16135463
- [Result] Nabid A, Choy H, Stea BD, et al.: Encouraging survival results with RSR13 and concurrent radiation therapy: interim analysis of a phase II study for locally advanced unresectable non-small cell lung cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1236, 2002.